CLINICAL TRIAL: NCT03439267
Title: Effectiveness of a Proactive Cardiovascular Primary Prevention Strategy, With or Without the Use of Coronary Calcium Screening, in Preventing Future Major Adverse Cardiac Events
Acronym: CorCal
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1050633
Record Dates: First submitted 2018-02-14; First posted 2018-02-20 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-01

CONDITIONS: Cardiovascular Primary Prevention Strategy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Proactive Current National Guidelines Group (Active Comparator): Standard Interventional Control Group. Will receive treatment recommendation according to the current National guidelines for statin initiation and follow-up.
  Interventions: Other: Standard Treatment
- Proactive CAC Group (Experimental): Investigational Interventional Group. Will undergo coronary artery calcium screening and will receive statin recommendation based on the cardiovascular risk algorithm.
  Interventions: Combination Product: Coronary Artery Calcium Screening and Statin Treatment

INTERVENTIONS:
Combination Product: Coronary Artery Calcium Screening and Statin Treatment — Will undergo coronary artery calcium screening and will receive statin treatment based on the cardiovascular risk algorithm.
  Arms: Proactive CAC Group
Other: Standard Treatment — Patients will be managed following the AHA/ACC guidelines for statin initiation and follow-up.
  Arms: Proactive Current National Guidelines Group

SUMMARY:
The primary objective of this study is to test the effectiveness of a proactive cardiovascular primary prevention strategy, with or without the use of coronary calcium screening, compared to current standard care, in preventing future major adverse cardiac events (MACE), including all-cause death, non-fatal myocardial infarction (MI), stroke, or any arterial revascularization among a moderate risk population with no current evidence of cardiovascular disease.

DETAILED DESCRIPTION:
This is a randomized, open-label, pragmatic study designed to assess the effectiveness of coronary calcium screening. Patients who provide consent, and are eligible, will be randomized 1:1 to receive statin recommendation based on coronary calcium screening results or standard risk assessment results using the American Heart Association/American College of Cardiology (AHA/ACC)-recommended pooled cohort equation.

Management of all participants will be done through their primary care physicians/clinicians and their qualified delegates who will receive education and training from the Principal Investigator and/or his delegate about the two treatment strategies. The current National guidelines group will be managed following the AHA/ACC guidelines for statin initiation and follow-up. The coronary artery calcium (CAC) group will undergo coronary artery calcium screening and will receive a statin recommendation based on the proposed CAC cardiovascular (CV) risk algorithm. All subjects will be asked to complete the Intermountain Statin Adherence Questionnaire (ISAQ) at 3 months after recommendation (+ 60 days) and then annually thereafter (within +/- 60 days of the anniversary date of recommendation). All subjects will remain under the usual care of their primary care physicians and will be followed by the study team via their electronic health records (EHR) for approximately an average of 4 years following the subjects' anniversary date of recommendation, but until the target primary endpoint event rate is met. All enrolled subjects will be followed for outcomes and this will be completely done by electronic medical records query. Other than the time point to obtain agreement for study participation and to perform the CAC screening and/or lipid panel, there will be no other study-specific clinic visits required. Further, there will be no other treatments or procedures required for this study. After about the first 600 patients are enrolled, an interim meeting will occur to evaluate entry criteria and size to determine if any modifications to the protocol should occur.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects 50 to 80 years of age or female subjects 60 to 80 years of age, of any ethnic origin
2. Ability to understand and provide agreement to study participation, which must be obtained prior to initiation of any study procedures
3. No known history, as documented in the EHR, of coronary artery disease, cerebrovascular disease, peripheral vascular disease, or diabetes mellitus at enrollment
4. Willing and able to provide access to their EHR until study end
5. Willing and able to undergo a computed tomography (CT) coronary artery calcium screening test
6. Current and/or past patients seen at Intermountain facilities and who have accessible EHR at the facility(ties) where they are seen.

Exclusion Criteria:

1. Patients who have active on-going cancer or are on dialysis
2. Any evidence of statin use prior to study participation
3. Participation in any other clinical trials involving investigational or marketed products within 30 days prior to entry in the study
4. Any evidence of a CAC test within the last 5 years prior to screening
5. The Study Doctor(s) determine(s) that the subject is not eligible for participation in this research study
6. The subject is non-English speaking, and therefore may be unable to fully understand the written and spoken instructions that may relate to the proper conduct of the trial

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5765 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
MACE | 5 years
  Composite of all-cause mortality, myocardial infarction, stroke, and revascularization (coronary, carotid, and peripheral).

CONTACTS AND LOCATIONS:
Overall Officials: Joseph B Muhlestein, MD, Principal Investigator — Intermountain Medical Center
Locations (1):
- Intermountain Medical Center and Intermountain Clinics, Murray, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Muhlestein JB, Knowlton KU, Le VT, Lappe DL, May HT, Min DB, Johnson KM, Cripps ST, Schwab LH, Braun SB, Bair TL, Anderson JL. Coronary Artery Calcium Versus Pooled Cohort Equations Score for Primary Prevention Guidance: Randomized Feasibility Trial. JACC Cardiovasc Imaging. 2022 May;15(5):843-855. doi: 10.1016/j.jcmg.2021.11.006. Epub 2021 Dec 15. PMID 34922872